| Men Engagement in Women Empowerment for Improving Materi | nal |
|--------------------------------------------------------------|-----|
| Mental Health through Cash Transfer and Life Skills Building | |

MEWE (Men Engagement in Women Empowerment)

NCT Number: **04125251** 

Date of the Document: 19th July, 2019

#### **Informed Consent**

| Project title: | Project number: |
|---|---|
| Men Engagement in Women Empowerment | 51625 |
| for Improving Maternal Mental Health through | |
| Cash Transfer and Life Skills Building | |
| ERC Ref. No. 2019-1210-3832 | <b>Sponsor:</b> Bill and Melinda Gates Foundation |
| Principal Investigator: | Organization: |
| Dr. Zulfiqar Bhutta | Aga Khan University, Centre of Excellence in Women and |
| | Child Health (AKU-COE-WCH) |
| Location: | Phone: |
| Karachi, Pakistan | 021-34864724 |
| Other Investigators: | Organization: |
| Co-Lead: | |
| Dr. Rozina Karmaliani | Aga Khan University, School of Nursing and Midwifery |
| Dr. Tazeen Saeed Ali | Aga Khan University, School of Nursing and Midwifery |
| Technical Advisor: | |
| Dr. Judith McFarlane | Texas Women's University, Houston USA |
| Co-investigators: | |
| Dr. Saima Hirani | Aga Khan University, School of Nursing and Midwifery |
| Ms. Shireen Shehzad | Aga Khan University, School of Nursing and Midwifery |
| Dr. Nargis Asad | Aga Khan University, Department of Psychiatry |
| Mr. Hussain Maqbool Khuwaja | Aga Khan University, School of Nursing and Midwifery |
| Project Staff: | |
| Dr. Nasim Zahid Shah | AKU-COE-WCH |
| Mr. Zahid Hyder Khuwaja | AKU-COE-WCH |
| Mr. Shiraz Lalani | AKU-COE-WCH |
| Location: | Phone: |
| Karachi, Pakistan | 0213486-5461, 0213486-5480 |

I am \_\_\_\_\_ from Aga Khan University, Centre of Excellence in Women and Child Health (AKU-COE-WCH). The department is conducting a research on issues related to maternal and child health in Pakistan.

## **PURPOSE OF THE RESEARCH STUDY:**

This study addresses the psychosocial issues confronting women depression, domestic violence and simultaneously enhances the psychological functioning of women and children. Literature review on women health indicates a strong contrary association between depressions, domestic violence, economic deprivation and unfavorable health outcome for women and children. The Aga Khan University, in collaboration with Benazir Income Support Program (BISP), would intent to undertake a randomized controlled trial to train/teach and share information with the BISP beneficiary women along with their spouses regarding essential Life Skills Building (LSB) concepts in order to bring family harmony and healthy home environment.

## **PROCEDURES:**

Your participation in the project will require you/your spouse to give 2-3 hours per week for 10-12 weeks (2-3 months) in LSB training sessions.

# Life Skill Building Training among Cash Transfer beneficiaries and their spouse of Benazir Income Support Program (BISP)

There are altogether 10 modules based on different skills required for managing their daily routine. The skills included in the modules are communication skills, understanding roles of men and women, work life balance and time management, conflict resolution, dealing with abuse and harassment, enhancing self-efficacy, effective parenting and money management skills. If you/your spouse agree to be the participant for this study and your/your spouse name gets selected for this intervention then you and your spouse will be expected to attend 2-3 hour session per week. The training will be conducted in separate male and female groups, facilitated by master trainers on your convenient timing.

Before and after intervention you and your spouse will be expected to fill below mentioned forms for assessment, which will be collected by another data collector. The assessment forms will measure your mental health. The forms will require 50-60 minutes for completion. You/your spouse will be given help to fill the forms. The details of the forms are given above.

The brief details of the questioners are as follow:

- 1. **Demography** (In this form you will ask to fill about the basic demographic information about you and your family that also include question about work, income/economic solvency and housing characteristics, it will require 5-8 minutes).
- 2. **General Self-Efficacy Scale (GSE)** (In this you will be showing your coping and ability to deal with difficulties, this form will require 3-5 minutes).
- 3. **The Revised Conflicts Tactics Scales (CTS2S)** (You will asked about concerns related to household quarrels, it will require your 3-5 minutes).
- 4. **Patient Health Questionnaire (PHQ-9)** (This form will find out your responses towards various problems, it will need your 5 minutes).
- 5. Six-item Food Security Questionnaire (FSQ) (It will require your 5-10 minutes)
- 6. Gender Equitable Attitude Scale (GEAS) (it will require 5-8 minutes).
- 7. **Resilience Scale** (it will require 5-8 minutes)

#### **CONFIDENTIALITY:**

Data will be collected in a separate room. We assure you/your spouse that all the information gathered will be kept confidential by using unique participants' identification number instead of name. Only authorized researchers will have the access to the information. Even your family will not have right to use your information. Any published material coming out of this study will not use your/your spouse name. However, Ethics Review Committee (ERC) at Aga Khan University or any regulatory body can have direct access to your data for monitoring and audit.

## **POSSIBLE BENEFITS:**

If the need of professional help is identified, regarding mental illnesses, Dr. Nargis Asad (clinical Psychologist) will provide consultation or referral, if needed. Your referral will be kept confidential. Your early identification will ensure better prognosis.

#### POSSIBLE RISKS OR DISCOMFORT:

You may find items on the form personal and could feel some discomfort while answering them. You may choose not to answer any or all questions. Your participation in this research will not have any effect on your monthly cash transfer from BISP.

## **WITHDRAWAL WITHOUT PREJUDICE:**

You may choose to withdraw from this study at any time. There is no penalty for withdrawing from the study. It will not have any effect on the services available to you. Participating in this study is on voluntarily basis.

## FINANCIAL CONSIDERATION:

You do not have to pay for taking part in this study. Similarly, Your will not get money to be part of this study but will be getting refreshment during the LSB training.

## **AVAILABLE SOURCES OF INFORMATION:**

If there are any questions about the research, Dr. Rozina Karmaliani, Dr. Tazeen Saeed Ali and Dr. Nargis Asad will be happy to respond. You could contact them at the Aga Khan University, School of Nursing, in Karachi. Their phone numbers are 21-3486-5461, or 21-3486-5480, or 21-3486-4699, respectively.

This study has been reviewed and approved by AKU- ERC. If you have any question regarding your legal rights, you may contact at 021-3486-4880

## **AUTHORIZATION:**

I have read this consent form and my questions have been answered. By signing this consent form I will not give up any of my legal rights. I will be given a signed copy of this consent form.

| Name of Participant | | Signature of Participant | Date |
|---|---|---|---|
| or<br>Name of Participant's Legal<br>Acceptable Representative | or | Signature of Participant's<br>Legal Acceptable<br>Representative | Date |
| If illiterate. | | | |

| Witness: | | |
|---|---|---|
| | of the consent form to the potential parti<br>sk questions. I confirm that the individu | • |
| Name and signature of witness: | Date: | |
| Printed Name of Person<br>Obtaining Consent | Signature of Person Obtaining<br>Consent | Date |
| Name of Principal Investigator | Signature of Principal Investigator | Date |